CLINICAL TRIAL: NCT05028556
Title: A Phase 1, Multicenter, Open-label, Dose-increasing Study to Evaluate the Safety, Tolerability, PK/PD and Preliminary Efficacy of Y101D, a Recombinant Anti-PD-L1 and TGF-β Bispecific Antibody for Injection, in Patients With Metastatic or Locally Advanced Solid Tumors
Brief Title: A Trial of Y101D, a PD-L1/TGF-β Bispecific Antibody, in Patients With Metastatic or Locally Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wuhan YZY Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y101D01
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Metastatic or Locally Advanced Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Y101D (Experimental): Y101D in subjects with Metastatic or Locally Advanced Solid Tumors
  Interventions: Drug: Cohort 1 of Y101D; Drug: Cohort 2 of Y101D; Drug: Cohort 3 of Y101D; Drug: Cohort 4 of Y101D; Drug: Cohort 5 of Y101D

INTERVENTIONS:
Drug: Cohort 1 of Y101D — Y101D, 1mg/kg, Q2W, intravenous infusion
Drug: Cohort 2 of Y101D — Y101D, 3mg/kg, Q2W, intravenous infusion
Drug: Cohort 3 of Y101D — Y101D, 10mg/kg, Q2W, intravenous infusion
Drug: Cohort 4 of Y101D — Y101D, 20mg/kg, Q2W, intravenous infusion
Drug: Cohort 5 of Y101D — Y101D, 30mg/kg, Q2W, intravenous infusion

SUMMARY:
This is a phase 1, multicenter, open-label study to evaluate the safety, tolerability, PK, PD, immunogenicity and preliminary efficacy of Y101D in patients with metastatic or locally advanced solid tumors.

DETAILED DESCRIPTION:
This study will consist of two parts: dose escalation part and cohort expansion part.

In dose escalation part, up to 5 dose-escalation cohorts will be sequentially enrolled in this study. The five dose levels are 1, 3, 10, 20 and 30 mg/kg. DLTs will be evaluated during the first treatment cycle, which is 28 days. The study consists of a 4-week screening period, a 4-week core treatment period for DLT evaluation, a treatment extension period, a safety follow-up visit for approximately 30 days following the last dose of Y101D, and survival follow-ups every 3 months thereafter.

In cohort expansion part, To further characterize safety and efficacy of Y101D, cohort expansion will be allowed in the following two circumstances: MTD cohort expansion if the MTD could be identified; Benefited dose cohort if it could be determined by Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 (including 18 and 75 years old), gender is not limited;
2. Pathologically confirmed metastatic or locally advanced solid tumors with failure or absence of standard care;
3. ECOG physical status score must be 0~1;
4. Expected survival of subjects evaluated by the investigator ≥3 months;
5. Hemogram: absolute neutrophil count (ANC) ≥1.5×109/L, hemoglobin ≥90g/L (no red blood cells were injected within 14 days before the first administration), platelet ≥90×109/L;
6. Liver: bilirubin ≤1.5 times the upper limit of normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal value;If the subject has liver metastasis, ALT and AST are allowed to be less than 5 times the upper limit of normal value;
7. Kidney: Serum creatinine ≤1.5 times the upper limit of normal value or creatinine clearance ≥ 60 mL/min (using standard Cockcroft-Gault formula);
8. Understand and voluntarily sign written informed consent.

Exclusion Criteria:

1. Have received chemotherapy, radiotherapy (local palliative radiotherapy for 14 days) and immunotherapy within 28 days before the first administration, and have received small molecule targeted drugs or Chinese patent drugs with anti-tumor indications within 14 days;
2. Major surgery (except diagnostic biopsy) within 28 days prior to the first dose;
3. Subjects with central nervous system (CNS) metastases causing clinical symptoms or requiring therapeutic intervention;Patients who had previously received BMs were included if they were asymptomatic ≥4 weeks prior to initial dosing, had stable disease on radiographic findings, and did not require corticosteroid or anticonvulsant therapy;
4. Receive any organ transplantation, including allogeneic stem cell transplantation, except those that do not require immunosuppression (e.g. cornea transplantation, hair transplantation);
5. Adverse events caused by previous antitumor therapy have not recovered (i.e., grade 1 or at baseline), except for hair loss and grade 2 neuropathy, hormone replacement hypothyroidism, or other confirmed chronic adverse events;
6. Subjects with a history of malignancy (non-study tumor) within 3 years prior to the first study administration date (other than skin squamous cell carcinoma and basal cell carcinoma, carcinoma in situ of the cervix or breast, or other non-invasive lesions that the Investigator and Sponsor agree have been cured and have a very low risk of recurrence within 3 years);
7. Have a known allergy, hypersensitivity or intolerance to corticosteroids, monoclonal antibodies or human proteins or their excipients;
8. Uncontrolled active infection (CTCAE≥2);
9. Subjects with severe respiratory diseases judged by the researcher to be unsuitable for inclusion;
10. Subjects with a history of serious cardiovascular disease, including previous coronary artery bypass grafting or stent implantation, myocardial infarction or cerebrovascular accident within 6 months, history of congestive heart failure or unstable angina pectoris, uncontrolled severe hypertension, and arrhythmias requiring medication;
11. Active autoimmune diseases (such as inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus (sle), hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis, etc.), into the group when the disease is in stable except ZhuangTaiZhe (no need to systemic immune inhibitors to treat symptoms stable under the condition of more than 6 months).
12. Subjects with uncontrolled metabolic diseases such as diabetes, severe gastrointestinal bleeding, and severe diarrhea (CTCAE≥2), and subjects with severe gastrointestinal obstruction requiring intervention;
13. Human immunodeficiency virus (HIV) antibody positive, hepatitis B virus (HBV) surface antigen positive and HBV DNA test indicated active hepatitis B (HBV-DNA≥1000cps/ml), active hepatitis C (hepatitis C antibody positive and HCV-RNA higher than the detection limit of the analysis method), active syphilis;
14. Those who received live (attenuated) virus vaccine within 4 weeks before the first administration;
15. Pregnant or lactating women or men or women who have a birth plan within 12 months;
16. Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia;
17. Subjects with poor compliance or who are considered by the Investigator to be unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | From the time of the first dose (Day 1) until the 2nd dosing (Day 28)
  DLTs were assessed using the national cancer institute common terminology criteria for adverse events (NCI-CTCAE) version 5.0.
Adverse Events according to CTCAE V5.0 | Time Frame: From the start of administration to the end of the study or 28 days after the administration is stopped (up to 6 months and 28 days)
  An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Area under the curve (AUC) of Y101D | Up to 1 weeks after the 2nd dosing
Peak Plasma Concentration (Cmax) of Y101D | Up to 1 weeks after the 2nd dosing
Half-time (t1/2) of Y101D | Up to 1 weeks after the 2nd dosing
immunogenicity | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The presence of antibodies directed against the biotherapeutic medicine upon administration, including the ADA and Nab.
Objective Response Rate (ORR) | 6 months (anticipated)
  ORR is defined as percentage of participants who achieved complete response (CR), partial response (PR), based on RESIST 1.1.
Time to Progression (TTP) | 6 months (anticipated)
  TTP was defined as the number of days from the date of first infusion (Day 1) to the date of first record of disease progression.
Duration of Response | 6 months (anticipated)
  Duration of response was calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in RESIST 1.1.
Progression-Free Survival (PFS) | 6 months (anticipated)
  PFS was defined as the time between the date of first dose of Y101 and either disease progression or death, whichever occurs first.
Overall Survival (OS) | 12 months (anticipated)
  OS was defined as the number of days from administration of the first infusion (Day 1) to date of death.
Time to first Response | 6 months (anticipated)
  Time to first response was defined as the time from the date of first dose of Y101 to the date of initial documentation of a response (PR or better).

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Cancer Prevention Center, Sun Yat-sen University
Locations (3):
- China (3):
  - Cancer Prevention Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No